CLINICAL TRIAL: NCT02575547
Title: Effect of Neoadjuvant Chemotherapy Followed by Concurrent Chemo-radiotherapy on Nutritional Status in Locoregionally Advanced Nasopharyngeal Carcinoma Patients: Prospective Observational Study
Brief Title: Effect of Chemoradiotherapy on Nutritional Status in Advanced NPC Patients
Status: Completed | Type: Observational
Sponsor: Zhao Chong (Other)
Collaborators: Wuhan University (Other); Fudan University (Other); Fujian Cancer Hospital (Other Government); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Cancer Hospital of Guizhou Province (Other); Hainan People's Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Sponsor-Investigator, Zhao Chong, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2015-FXY-034-Nutrition and NPC
Record Dates: First submitted 2015-09-19; First posted 2015-10-14 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Nasopharyngeal Carcinoma; Malnutrition
Keywords: Nutritional Status; Locoregionally Advanced Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Malnutrition | interventions — Cisplatin; Docetaxel; Radiation; Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NC+CCRT: Patients treated with neoadjuvant chemotherapy(NC) (cisplatin and docetaxel) and CCRT (cisplatin)
  Interventions: Drug: cisplatin and docetaxel

INTERVENTIONS:
Drug: cisplatin and docetaxel — NC：cisplatin 75 mg/m2 intravenous infusion in day1，docetaxel 75 mg/m2 intravenous infusion in day1，both drugs are given every 3 weeks, two courses.
  CCRT: intensity modulation radiation therapy(IMRT) and cisplatin (100mg/m2 on day 1) every three weeks for three\three cycles during radiation therapy(RT).
  Dietary supplement: enteral nutrition and parenteral nutrition
  Other Names: radiation; enteral nutrition and parenteral nutrition

SUMMARY:
This is an prospective，open-label, none-interventional, observational， multicenter phase II clinical trial. The purpose of this study is to observe the effect of neoadjuvant chemotherapy followed by concurrent chemoradiation therapy(CCRT) on nutritional status in locoregionally advanced nasopharyngeal carcinoma(NPC) patients, analyse the changes of patients' nutrition status during the treatment and the connection between nutrition changes and curative effects, evaluate nutritional risks under the neoadjuvant chemotherapy and CCRT and provide data and basis for further study。

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma(WHO II)
* All genders，range from 18～65 years old
* Karnofsky performance status(KPS) ≥ 80
* Clinical stage III~IVb(UICC 7th)
* Without significant digestive system disease，nutritional and metabolic diseases or endocrine disease
* Without significant cardiac，respiratory，kidney or liver disease
* Not received radiotherapy, chemotherapy and other anti-tumor treatment(including immunotherapy)
* white blood cell(WBC) count ≥ 4×109/L, neutrophile granulocyte(NE) count ≥ 1.5×109/L, Hemoglobin(HGB) ≥ 10g/L, platelet(PLT) count ≥ 100×109/L
* alanine aminotransferase (ALT) or aspartate aminotransferase(AST) < 1.5×upper limit of normal(ULN), bilirubin < 1.5×ULN, alanine aminotransferase (CCR) ≥ 30ml/min
* Inform consent form

Exclusion Criteria:

* Distance metastases
* Second malignancy within 5 years
* Drug or alcohol addition
* Do not have full capacity for civil acts
* Active systemic infections
* Chronic consumptions
* Mental disorder
* Pregnancy or lactation
* Concurrent immunotherapy or hormone therapy for other diseases
* Severe complication, eg, uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: III-IVb(Union for International Cancer Control,UICC 7th) NPC patients with histologic diagnosis of World Health Organization(WHO) II
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in Body weight | baseline and 36 months

SECONDARY OUTCOMES:
Acute Toxicity | 3 months
  To evaluate the acute toxicity with Common Terminology Criteria For Adverse Events (CTCAE) 3.0 when adjuvant chemotherapy and concurrent chemoradiation is used.
Number of Participants With Abnormal Laboratory Values | 36 months
  To observe patients' complete blood cell count and blood biochemical examination during the treatment and three years after the treatment.
Adverse Events That Are Related to Treatment | 36 months
  Using European Organization for Research and Treatment of Cancer(EORTC) quality of life questionnaire(QLQ)-C30(version 3.0) and EORTC QLQ-H&N35(Version 1.0) to access the quality of life. Collecting data before treatment, 1 week after each 4/5 cycles of chemotherapy, 3 years after all treatment finished.
Tumor regressive rate after treatment | 36 months
Late toxicity | 36 months
  To evaluate the late toxicity with the SOMA criterion after 1/2/3 years of treatment.
Three-year locoregional relapse free survival rate | 36 months
Three-year distance metastasis free survival rate | 36 months
Three-year overall survival rate | 36 months
Three-year disease free survival rate | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Miao J, Wang L, Ong EHW, Hu C, Lin S, Chen X, Chen Y, Zhong Y, Jin F, Lin Q, Lin S, Hu X, Zhang N, Wang R, Wang C, Guo X, Yit NLF, Shi H, Tan SH, Mai H, Xie C, Chua MLK, Zhao C. Effects of induction chemotherapy on nutrition status in locally advanced nasopharyngeal carcinoma: a multicentre prospective study. J Cachexia Sarcopenia Muscle. 2023 Apr;14(2):815-825. doi: 10.1002/jcsm.13196. Epub 2023 Mar 5. PMID 36872457
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn